CLINICAL TRIAL: NCT05951660
Title: The Effect of Targeted Education on Number, Severity, and Perception of Sexual Side Effects of Patients Suffering From Schizophrenia and Diabetes or Prediabetes.
Brief Title: Sex, Psychopharmacology, and Diabetes
Acronym: SECRET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Steno Diabetes Center Sjaelland (Other Government); University College Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EMN-2022-08015, SJ-1005
Record Dates: First submitted 2023-07-10; First posted 2023-07-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Diabetes Mellitus; PreDiabetes; Sexual Dysfunction; Drug-Related Side Effects and Adverse Reactions; Education
Keywords: Randomized Controlled Trial; Treatment Adherence and Compliance; Antipsychotic Agents; Patient Education as Topic
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Diabetes Mellitus; Prediabetic State; Sexual Dysfunction, Physiological; Drug-Related Side Effects and Adverse Reactions; Treatment Adherence and Compliance | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- INT1: Only patients are educated (Experimental)
  Interventions: Behavioral: Educational intervention
- INT2: Only Healthcare Professionals are educated (Experimental)
  Interventions: Behavioral: Educational intervention
- INT3: Both patients and Healthcare Professionals are educated (Experimental)
  Interventions: Behavioral: Educational intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Educational intervention — Different teaching sessions are used for patients and healthcare professionals, respectively.
  The teaching sessions are held at the Assertive Community Treatment (ACT) Centers from which the patients are recruited. The duration is 3x30 minutes with breaks for patients and 60 minutes for healthcare professionals. Teaching sessions are held by two doctors a specialist in clinical pharmacology and a specialist in psychiatry and clinical sexology providing the participants with knowledge and tools for the dialogue on SD and drug-related side effects.
  The topics of the teaching sessions are:
  * What is sexuality?
  * How psychopharmacology influences sexuality
  * What can be done?
  The topics will be addressed in a mixture of short informative talks using a PowerPoint presentation, group discussions, and exchanges of personal experiences.
  Arms: INT1: Only patients are educated; INT2: Only Healthcare Professionals are educated; INT3: Both patients and Healthcare Professionals are educated

SUMMARY:
The term sexual (SD) dysfunction covers conditions that prevent people from having a satisfactory sex life. SD is a frequent and sometimes debilitating complication of mental illness and a known adverse reaction to psycho-pharmacological treatment. SD is also associated with diabetes, a common somatic comorbidity in psychiatric patients. SD is associated with both reduced quality-of-life and reduced treatment adherence, yet SD is far too rarely addressed between the patient and the healthcare professional in clinical consultations.

The purpose of the study is to investigate whether targeted education of patients with schizophrenia and diabetes/prediabetes and/or their healthcare professionals in causes and management of SD:

* Increases the number of systematic examinations of sexual side effects,
* Causes changes in the psycho-pharmacological treatment, and
* Reduces the severity or perception of sexual side effects.

The study is a multicenter Randomized Controlled Trial (RCT) with four arms, in which the educational intervention is provided to patients, healthcare professionals, or both groups. The effect of the educational intervention is compared to a non-educated control group. The study is expected to include 192 patients recruited from 16 assertive community treatment centers evenly distributed in four Danish regions.

The study is part of an interdisciplinary project named SECRET. The educational intervention was developed in an ethnographic pre-study incorporating stakeholder engagement. Parallel to the present RCT, an ethnographic field study will be carried out to broaden the perspective on the effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A diagnosis in the schizophrenic spectrum (ICD10 F2x)
* One of the following:

  1. A diagnosis of diabetes (ICD10 E10x, E11x, E12x, E13x, 14x)
  2. A current or previous prediabetes defined as an HbA1c between 39-47 mmol/mol (both included) measured in at least two blood samples collected with ≥3 months intervals as part of the patient's routine clinical monitoring
  3. Obesity defined as a Body-Mass Index (BMI) ≥30 kg/m2
* Ongoing treatment with at least one antipsychotic agent
* A SD that can be rated using Changes in Sexual Function Questionnaire-14 (CSFQ-14)

Exclusion Criteria:

* Incapacitated or subject to mental health probation
* Unable to speak danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to follow up in the total score of Changes in Sexual Function Questionnaire-14 (CSFQ-14) | At inclusion and at follow-up, i.e. 6 months after the educational intervention is finished.
  Measured by Changes in Sexual Function Questionnaire-14 (CSFQ-14)

SECONDARY OUTCOMES:
Changes in psycho-pharmacological treatment | Recorded continuously throughout the entire study period, i.e. from the day of the educational intervention to 6 months after the end of the educational intervention.
  Estimated by changes in prescribed medications
The frequency in which sexual issues are discussed in the clinical consultation | Recorded continuously throughout the entire study period, i.e. from the day of the educational intervention to 6 months after the end of the educational intervention.
  The number of systematic examinations of sexual side effects estimated by the number of consultations where sexual side effects are addressed, and whether it is the patient or the healthcare professional, who addresses the subject.
Changes from baseline to follow up in compliance / Adherence to the Pharmacological Treatment | At inclusion and at follow-up, i.e. 6 months after the educational intervention is finished.
  Measured by Rating of Medication Influences (ROMI) Scale
Changes from baseline to follow up in shared decision making | At inclusion and at follow-up, i.e. 6 months after the educational intervention is finished.
  Measured by Shared Decision Making-9 (SDM) measurement tool

CONTACTS AND LOCATIONS:
Overall Officials: Gesche Jürgens, Clinical Professor, Study Chair — Clinical Pharmacology Unit, Zealand University Hospital, Roskilde, Denmark; Annamaria Giraldi, Clinical Professor, Principal Investigator — Sexological Clinic, Psychiatric Centre Copenhagen, Denmark; Lise Tarnow, MD, DMSc, Principal Investigator — Steno Diabetes Center Sjaelland, Denmark; Charlotte Bredahl Jacobsen, Senior Researcher, PhD., Principal Investigator — Institute of Social Work, University College Copenhagen, Copenhagen, Denmark; Rikke Meyer, MD, Principal Investigator — Clinical Pharmacology Unit, Zealand University Hospital, Roskilde, Denmark
Locations (1):
- Assertive Community Centres, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No